CLINICAL TRIAL: NCT00243204
Title: Study of Talabostat + Docetaxel Versus Docetaxel in Stage IIIB/IV Non-Small Cell Lung Cancer (NSCLC) After Failure of Platinum-Based Chemotherapy
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: FDA Hold May 2007
Sponsor: Point Therapeutics (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PTH-304
Record Dates: First submitted 2005-10-19; First posted 2005-10-21 (Estimated); Last update posted 2007-06-08 (Estimated); Status verified 2007-06

CONDITIONS: Carcinoma, Non-Small Cell Lung
Keywords: Stage IIIb/IV non-small cell lung cancer; NSCLC; Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms | interventions — PT-100 dipeptide; Docetaxel

INTERVENTIONS:
Drug: talabostat mesylate
Drug: docetaxel

SUMMARY:
This Phase 3 study will compare the efficacy of talabostat plus docetaxel to docetaxel plus placebo in patients with Stage IIIB/IV NSCLC who have failed a platinum-based chemotherapy regimen.

ELIGIBILITY:
INCLUSION CRITERIA:

* Men or women age 18 years or older
* Histologically or cytologically confirmed NSCLC

  * Recurrent, locally advanced or metastatic, inoperable NSCLC (Stage IIIB/IV)
  * Patients with Stage IIIB NSCLC must have a cytologically documented pleural effusion
* Failed or relapsed after receiving a platinum-containing chemotherapy regimen as first-line therapy for advanced NSCLC
* Measurable disease on computerized tomography (CT) scan
* ECOG Performance Status of 0 or 1
* Expected survival ≥12 weeks
* Provide written informed consent

EXCLUSION CRITERIA:

* More than 2 prior chemotherapy regimens
* Clinically significant laboratory abnormalities, specifically:

  * Total bilirubin ≥ institutional upper limit of normal (ULN)
  * Serum alanine aminotransferase (ALT) or aspartate aminotransferase (AST) ≥1.5 x ULN concomitant with alkaline phosphatase >2.5 x ULN
  * Serum creatinine ≥2.0mg/dL
  * Absolute neutrophil count <1500/μL or platelets <100,000/μL
* Untreated or symptomatic brain metastases
* Any malignancy within the 5 years immediately prior to the first dose of study medication with the exception of basal cell or non-metastatic squamous cell carcinoma of the skin, and carcinoma in-situ of the cervix
* A history of severe hypersensitivity to drugs formulated with polysorbate 80
* Any comorbidity or condition which, in the opinion of the investigator, may interfere with the assessments and procedures of this protocol
* Patients who are within 28 days of chemotherapy, radiation therapy, immunotherapy, or other investigational medication for NSCLC.
* Pregnancy or lactation. Women of childbearing potential and non-vasectomized men must agree to use a barrier method of contraception.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2006-01

CONTACTS AND LOCATIONS:
Locations (96):
- United States (96):
  - Marshall Schreeder, MD, Huntsville, Alabama
  - James P. Daugherty, MD, Muscle Shoals, Alabama
  - Alaska Cancer Research, Anchorage, Alaska
  - Hematology Oncology Associates, Phoenix, Arizona
  - Veena Charu, MD, Anaheim, California
  - Lalita Pandit, MD, Inc, Fountain Valley, California
  - Robert A. Moss, MD, FACP, Inc., Fountain Valley, California
  - Warren Paroly, MD, Oceanside, California
  - Swarna S. Chanduri, MD, Pomona, California
  - Southwest Cancer Care Medical Group, Poway, California
  - Mile High Oncology, Denver, Colorado
  - Rocky Mountain Cancer Centers, Denver, Colorado
  - Medical Specialists of Fairfield, Fairfield, Connecticut
  - Pasco Hernando Oncology Associates PA, Brooksville, Florida
  - Lucio Gordan, MD, Gainesville, Florida
  - Citrus Hematology and Oncology Center, Inverness, Florida
  - Nature Coast Clinical Research, LLC, Inverness, Florida
  - Jorge G. Otoya, MD, Kissimmee, Florida
  - Cancer and Blood Disease Center, Lecanto, Florida
  - Pasco Hernando Oncology Associates, PA, New Port Richey, Florida
  - Ocala Oncology Center, Ocala, Florida
  - Cancer Center of Florida, Ocoee, Florida
  - Hematology Oncology Associates of Illinois, Chicago, Illinois
  - University of Chicago, Chicago, Illinois
  - Joliet Oncology Hematology Associates, Joliet, Illinois
  - Indiana Hematology Oncology Consultants, Indianapolis, Indiana
  - Northern Indiana Oncology Associates, South Bend, Indiana
  - Kansas City Cancer Centers, Southwest, Overland Park, Kansas
  - Kentucky Cancer Clinic, Hazard, Kentucky
  - Medical Oncology, LLC, Baton Rouge, Louisiana
  - Maryland Oncology Hematology, PA, Columbia, Maryland
  - Chesapeake Oncology Hematology Associates (Tate Center), Glen Burnie, Maryland
  - Josephine Ford Cancer Center -- Downriver, Brownstown, Michigan
  - Michael McKenzie, DO, Clinton Township, Michigan
  - Henry Ford Medical Center -- Fairlane, Dearborn, Michigan
  - Henry Ford Health System, Detroit, Michigan
  - Youssef Hanna, MD, Port Huron, Michigan
  - Cancer and Transplant Consultants, PLC, Rochester Hills, Michigan
  - Cancer Care Associates, Rochester Hills, Michigan
  - Cancer Care Associates, PC, Royal Oak, Michigan
  - Hematology Oncology Consultants, Royal Oak, Michigan
  - Jeffrey H. Margolis, MD, Royal Oak, Michigan
  - William Beaumont Hospital, Royal Oak, Michigan
  - Oncology Care Associates, PLLC, Saint Joseph, Michigan
  - Michigan Hematology and Oncology Institute, Southgate, Michigan
  - Mitchell Folbe, MD, PC, Troy, Michigan
  - William Beaumont Hospital, Troy, Michigan
  - Henry Ford Medical Center, West Bloomfield, Michigan
  - St. Joseph Oncology, Inc., Saint Joseph, Missouri
  - Arch Medical Services, Inc., St Louis, Missouri
  - Billings Clinic, Billings, Montana
  - Comprehensive Cancer Centers of Nevada, Las Vegas, Nevada
  - The Center for Cancer and Hematologic Disease, Cherry Hill, New Jersey
  - New York Oncology Hematology, PC, Albany, New York
  - George A. Zervos, MD, Glen Head, New York
  - Northwestern Carolina Oncology Hematology, Hickory, North Carolina
  - Gabrail Cancer Center, Canton, Ohio
  - Oncology/Hematology Care, Inc., Cincinnati, Ohio
  - Gabrail Cancer Center, Dover, Ohio
  - Dayton Hematology and Oncology, Kettering, Ohio
  - Mukesh C. Bhatt, MD, Medina, Ohio
  - Trilogy Cancer Center, Wooster, Ohio
  - Cancer Care Associates, Oklahoma City, Oklahoma
  - Cancer Care Associates, Tulsa, Oklahoma
  - Northwest Cancer Specialists, Northrup, Portland, Oregon
  - Shatish A. Shah, MD, Gettysburg, Pennsylvania
  - Medical Oncology Associates of Wyoming Valley, PC, Kingston, Pennsylvania
  - Rittenhouse Hematology Oncology Associates, Philadelphia, Pennsylvania
  - Chester County Hematology / Oncology Services, West Chester, Pennsylvania
  - Cancer Care Institute of Carolina, Aiken, South Carolina
  - Charleston Hematology Oncology, PA, Charleston, South Carolina
  - Palmetto Hematology Oncology, PC, Spartanburg, South Carolina
  - Texas Cancer Center, Arlington, Texas
  - Texas Oncology Cancer Center, Austin, Texas
  - Texas Cancer Center (Dallas Southwest), Dallas, Texas
  - Mary Crowley Medical Research Center, Dallas, Texas
  - Texas Cancer Center / Denton, Denton, Texas
  - El Paso Cancer Treatment Center, El Paso, Texas
  - Texas Oncology, PA, Fort Worth, Texas
  - US Oncology Research and Clinical Pharmacy, Fort Worth, Texas
  - Texas Cancer Center of Mesquite, Mesquite, Texas
  - Allison Cancer Center, Midland, Texas
  - West Texas Cancer Center, Odessa, Texas
  - Paris Regional Cancer Center, Paris, Texas
  - Texas Oncology Cancer Center--Sugar Land, Sugar Land, Texas
  - Annandale-Fairfax Virginia Hematology Oncology, PC, Fairfax, Virginia
  - Peninsula Cancer Institute, Gloucester, Virginia
  - Peninsula Cancer Institute, Newport News, Virginia
  - Virginia Oncology Associates, Norfolk, Virginia
  - Oncology & Hematology Associates of Southwest Virginia, Inc., Salem, Virginia
  - Peninsula Cancer Institute, Williamsburg, Virginia
  - Masoom Kandahari, MD, PC, Woodbridge, Virginia
  - Puget Sound Cancer Centers, Seattle, Washington
  - Jay L. Wittenkeller, MD, Spokane, Washington
  - Cancer Care Northwest Research, Spokane, Washington
  - Northwest Cancer Specialists, PC, Vancouver, Washington